CLINICAL TRIAL: NCT01897519
Title: A Phase 2b, Randomized, Double-Blind, Placebo Controlled, Safety and Efficacy Trial of Multiple Dosing Regimens of ABT-719 for the Prevention of Acute Kidney Injury in Subjects Undergoing High Risk Major Surgery
Brief Title: A Safety and Efficacy Trial of Multiple Dosing Regimens of ABT-719 for the Prevention of Acute Kidney Injury in Subjects Undergoing High Risk Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Topline results from study M13-796 showed an overall lack of efficacy. There were no safety concerns.
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: M13-958; 2012-005710-19 (EudraCT Number)
Record Dates: First submitted 2013-05-10; First posted 2013-07-12 (Estimated); Last update posted 2014-06-06 (Estimated); Status verified 2014-06

CONDITIONS: Cardiothoracic Surgery; Vascular Surgery
Keywords: High risk surgery; Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury | interventions — ABT 719

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm 1 lower dose ABT-719 (Experimental)
  Interventions: Drug: ABT-719
- Arm 2 intermediate dose ABT-719 (Experimental)
  Interventions: Drug: ABT-719
- Arm 3 high dose ABT-719 (Experimental)
  Interventions: Drug: ABT-719
- Arm 4 Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Placebo infusion
  Arms: Arm 4 Placebo
Drug: ABT-719 — Arm 1 lower dose, arm 2 intermediate dose, arm 3 high dose
  Arms: Arm 1 lower dose ABT-719; Arm 2 intermediate dose ABT-719; Arm 3 high dose ABT-719

SUMMARY:
This study will evaluate the safety and efficacy of ABT-719 in patients undergoing high risk major surgery.

ELIGIBILITY:
Inclusion Criteria:

- Patients undergoing high risk major surgery in subjects with cardiovascular disease who are at risk of AKI.

Exclusion Criteria:

* Ongoing or recent history of sepsis
* Has recent documented acute kidney injury.
* Subject is scheduled to have a total or partial nephrectomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2013-05; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Change in urine Neutrophil Gelatinase-Associated Lipocalin (NGAL) | Day 0 to Day 7
  Comparison between each ABT-719 dose group versus placebo in the mean maximal change from baseline in urine NGAL from Day 0 - Day 7.

SECONDARY OUTCOMES:
Proportion of subjects that develop composite event at 90 days post surgery | 90 Day
  Develop at least one of the composite events: death, needing renal replacement therapy during the 90-day post operative period, or having a greater than 25% reduction in estimated or measured glomerular filtration rate.
Proportion of subjects that develop a composite event at 60 days post surgery | 60 Days
  Develop at least one of the composite events: death, needing renal replacement therapy during the 60-day post operative period, or having a greater than 25% reduction in estimated or measured glomerular filtration rate.
Proportion of subjects that develop the Acute Kidney Injury Network (AKIN) scoring criteria | Day 7
Proportion of subjects that develop the Kidney Disease Improving Global Outcomes (KDIGO) scoring criteria | Day 7

CONTACTS AND LOCATIONS:
Overall Officials: Ann Eldred, MD, Study Director — AbbVie
Locations (23):
- United States (20):
  - Site Reference ID/Investigator# 96295, Gainesville, Florida
  - Site Reference ID/Investigator# 96778, Jacksonville, Florida
  - Site Reference ID/Investigator# 96301, Tampa, Florida
  - Site Reference ID/Investigator# 96302, Fort Wayne, Indiana
  - Site Reference ID/Investigator# 101961, Indianapolis, Indiana
  - Site Reference ID/Investigator# 103356, Boston, Massachusetts
  - Site Reference ID/Investigator# 96303, Boston, Massachusetts
  - Site Reference ID/Investigator# 96997, Grand Blanc, Michigan
  - Site Reference ID/Investigator# 97878, Petoskey, Michigan
  - Site Reference ID/Investigator# 99377, Royal Oak, Michigan
  - Site Reference ID/Investigator# 99317, West Orange, New Jersey
  - Site Reference ID/Investigator# 96996, New York, New York
  - Site Reference ID/Investigator# 96296, Durham, North Carolina
  - Site Reference ID/Investigator# 102020, Cleveland, Ohio
  - Site Reference ID/Investigator# 103355, Columbus, Ohio
  - Site Reference ID/Investigator# 97556, Pittsburgh, Pennsylvania
  - Site Reference ID/Investigator# 103316, Providence, Rhode Island
  - Site Reference ID/Investigator# 102019, Memphis, Tennessee
  - Site Reference ID/Investigator# 108255, Charlottesville, Virginia
  - Site Reference ID/Investigator# 96300, Milwaukee, Wisconsin
- Denmark (3):
  - Site Reference ID/Investigator# 105755, Aarhus N
  - Site Reference ID/Investigator# 105757, Kolding
  - Site Reference ID/Investigator# 105756, Odense C